CLINICAL TRIAL: NCT06441643
Title: A Phase II, Prospective, Two-Stage, Double-Masked, Randomized, Multi-Center, Controlled, Dose-Response Study Assessing the Safety and Ocular Hypotensive Efficacy of AR-17043 and PG043 (AR-17043/Latanoprost) Ophthalmic Solutions in Subjects With Elevated Intraocular Pressure
Brief Title: Next Generation Rocklatan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLR305-E001
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: Glaucoma; IOP
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — Latanoprost; Ophthalmic Solutions; netarsudil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- AR-17043 low concentration (Stage 1) (Experimental): AR-17043 Ophthalmic Solution, one drop in each eye in the morning on Day 1, followed by one drop in each eye in the evening on Days 2-7.
  Interventions: Drug: AR-17043 Ophthalmic Solution
- AR-17043 medium concentration (Stage 1) (Experimental): AR-17043 Ophthalmic Solution, one drop in each eye in the morning on Day 1, followed by one drop in each eye in the evening on Days 2-7.
  Interventions: Drug: AR-17043 Ophthalmic Solution
- AR-17043 high concentration (Stage 1) (Experimental): AR-17043 Ophthalmic Solution, one drop in each eye in the morning on Day 1, followed by one drop in each eye in the evening on Days 2-7.
  Interventions: Drug: AR-17043 Ophthalmic Solution
- AR-17043 vehicle (Stage 1) (Placebo Comparator): AR-17043 Vehicle, one drop in each eye in the morning on Day 1, followed by one drop in each eye in the evening on Days 2-7.
  Interventions: Drug: AR-17043 Vehicle
- Rhopressa (Stage 1) (Active Comparator): Netarsudil 0.02% Ophthalmic Solution, one drop in each eye in the morning on Day 1, followed by one drop in each eye in the evening on Days 2-7.
  Interventions: Drug: Netarsudil 0.02% Ophthalmic Solution
- PG043 low concentration (Stage 2) (Experimental): PG043 Ophthalmic Solution, one drop in each eye in the evening on Days 1-28.
  Interventions: Drug: PG043 Ophthalmic Solution
- PG043 high concentration (Stage 2) (Experimental): PG043 Ophthalmic Solution, one drop in each eye in the evening on Days 1-28.
  Interventions: Drug: PG043 Ophthalmic Solution
- AR-17043 high concentration (Stage 2) (Active Comparator): AR-17043 Ophthalmic Solution, one drop in each eye in the evening on Days 1-28.
  Interventions: Drug: AR-17043 Ophthalmic Solution
- Latanoprost (Stage 2) (Active Comparator): Latanoprost 0.005% Ophthalmic Solution, one drop in each eye in the evening on Days 1-28.
  Interventions: Drug: Latanoprost 0.005% Ophthalmic Solution
- Rocklatan (Stage 2) (Active Comparator): Netarsudil 0.02%/Latanoprost 0.005% Ophthalmic Solution, one drop in each eye in the evening on Days 1-28.
  Interventions: Drug: Netarsudil 0.02%/Latanoprost 0.005% Ophthalmic Solution

INTERVENTIONS:
Drug: AR-17043 Ophthalmic Solution — Investigational monotherapy supplied in three concentration levels: low, medium, high
  Arms: AR-17043 high concentration (Stage 1); AR-17043 high concentration (Stage 2); AR-17043 low concentration (Stage 1); AR-17043 medium concentration (Stage 1)
Drug: PG043 Ophthalmic Solution — Investigational fixed dose combination supplied in two concentration levels: low and high
  Arms: PG043 high concentration (Stage 2); PG043 low concentration (Stage 2)
Drug: Latanoprost 0.005% Ophthalmic Solution — Marketed monotherapy
  Other Names: Latanoprost
  Arms: Latanoprost (Stage 2)
Drug: Netarsudil 0.02% Ophthalmic Solution — Marketed monotherapy
  Other Names: Rhopressa®
  Arms: Rhopressa (Stage 1)
Drug: Netarsudil 0.02%/Latanoprost 0.005% Ophthalmic Solution — Marketed fixed dose combination
  Other Names: Rocklatan®
  Arms: Rocklatan (Stage 2)
Drug: AR-17043 Vehicle — Placebo comparator
  Arms: AR-17043 vehicle (Stage 1)

SUMMARY:
The purpose of this two-stage clinical trial is to assess the safety and hypotensive efficacy of AR-17043 and PG043 ophthalmic solutions in subjects with open-angle glaucoma (OAG) or ocular hypertension (OHT).

DETAILED DESCRIPTION:
During Stage 1, approximately 100 adult subjects with OAG or OHT will be randomized to 5 arms: 3 different concentrations of AR-17043, placebo comparator, or netarsudil 0.02% (Rhopressa®) for a treatment duration of 7 days.

During Stage 2, approximately 350 adult subjects with OAG or OHT will be randomized to 5 arms: low and high concentrations of PG043 (AR-17043/latanoprost 0.005%), AR-17043 high concentration, latanoprost, or netarsudil 0.02%/latanoprost 0.005% (Rocklatan®) for a treatment duration of 28 days.

ELIGIBILITY:
Stage 1 Key Inclusion Criteria;

* Diagnosis of OAG or OHT in both eyes.
* High unmedicated IOP measurements in the study eye as specified in the protocol.
* Corrected visual acuity equal to or better than +1.0 logMAR (Snellen equivalent equal to or better than 20/200) in the study eye.
* Other protocol-specified inclusion criteria may apply.

Stage 2 Key Inclusion Criteria:

* Diagnosis of OAG or OHT in both eyes.
* High unmedicated IOP measurements in the study eye as specified in the protocol.
* Corrected visual acuity equal to or better than +0.7 logMAR (Snellen equivalent equal to or better than 20/100) in the study eye.
* Other protocol-specified inclusion criteria may apply.

Stage 1 and Stage 2 Key Exclusion Criteria:

* Current use of more than 2 ocular hypotensive medications within 30 days (either eye).
* Intraocular pressure greater than 36 millimeters mercury (mmHg) at Screening.
* Glaucoma other than OAG.
* Previous glaucoma surgery.
* Any abnormality preventing reliable measurements.
* Unable to demonstrate proper eyedrop instillation.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
Mean diurnal IOP at Day 8 (Stage 1) | Day 8 (8:00, 10:00, 12:00, 16:00)
  Intraocular pressure (IOP) will be measured with a Goldmann tonometer. Diurnal IOP will be calculated as the average of the four measurements.
Mean diurnal IOP at Day 29 (Stage 2) | Day 29 (8:00, 10:00, 16:00)
  Intraocular pressure (IOP) will be measured with a Goldmann tonometer. Diurnal IOP will be calculated as the average of the three measurements.

SECONDARY OUTCOMES:
Mean IOP at each post-treatment timepoint (Stage 1) | Day 1 (8:00, 10:00, 12:00), Day 8 (8:00, 10:00, 12:00, 16:00)
  Intraocular pressure (IOP) will be measured with a Goldmann tonometer at each post-treatment timepoint.
Mean change from the diurnally adjusted baseline IOP at each post-treatment timepoint (Stage 1) | Baseline (8:00, 10:00, 12:00, 16:00), Day 1 (8:00, 10:00, 12:00), Day 8 (8:00, 10:00, 12:00, 16:00)
  Intraocular pressure (IOP) will be measured with a Goldmann tonometer at each post-treatment timepoint and compared to the time-relevant (corresponding) baseline measurement. Baseline is defined as the last visit prior to initiation of treatment.
Mean percent change from diurnally adjusted baseline IOP at each post-treatment timepoint (Stage 1) | Baseline (8:00, 10:00, 12:00, 16:00), Day 1 (8:00, 10:00, 12:00), Day 8 (8:00, 10:00, 12:00, 16:00)
  Intraocular pressure (IOP) will be measured with a Goldmann tonometer at each post-treatment timepoint and compared to the time-relevant (corresponding) baseline measurement. Baseline is defined as the last visit prior to initiation of treatment.
Mean change from baseline mean diurnal IOP at each post-treatment timepoint (Stage 1) | Baseline (8:00, 10:00, 12:00, 16:00), Day 1 (8:00, 10:00, 12:00), Day 8 (8:00, 10:00, 12:00, 16:00)
  Intraocular pressure (IOP) will be measured with a Goldmann tonometer. The baseline mean diurnal IOP will be calculated as the average of the four baseline measurements. Baseline is defined as the last visit prior to initiation of treatment.
Mean percent change from baseline mean diurnal IOP at each post-treatment timepoint (Stage 1) | Baseline (8:00, 10:00, 12:00, 16:00); Day 1 (8:00, 10:00, 12:00), Day 8 (8:00, 10:00, 12:00, 16:00)
  Intraocular pressure (IOP) will be measured with a Goldmann tonometer. The baseline mean diurnal IOP will be calculated as the average of the four baseline measurements. Baseline is defined as the last visit prior to initiation of treatment.
Mean IOP at each post-treatment timepoint (Stage 2) | Day 8 (8:00, 10:00, 16:00); Day 15 (8:00, 10:00, 16:00); Day 29 (8:00, 10:00, 16:00)
  Intraocular pressure (IOP) will be measured with a Goldmann tonometer at each post-treatment timepoint.
Mean change from the diurnally adjusted baseline IOP at each post-treatment timepoint (Stage 2) | Baseline (8:00, 10:00, 16:00); Day 8 (8:00, 10:00, 16:00); Day 15 (8:00, 10:00, 16:00); Day 29 (8:00, 10:00, 16:00)
  Intraocular pressure (IOP) will be measured with a Goldmann tonometer at each post-treatment timepoint and compared to the time-relevant (corresponding) baseline measurement. Baseline is defined as the last visit prior to initiation of treatment.
Mean percent change from diurnally adjusted baseline IOP at each post-treatment timepoint (Stage 2) | Baseline (8:00, 10:00, 16:00); Day 8 (8:00, 10:00, 16:00); Day 15 (8:00, 10:00, 16:00); Day 29 (8:00, 10:00, 16:00)
  Intraocular pressure (IOP) will be measured with a Goldmann tonometer at each post-treatment timepoint and compared to the time-relevant (corresponding) baseline measurement. Baseline is defined as the last visit prior to initiation of treatment.
Mean change from baseline mean diurnal IOP at each post-treatment timepoint (Stage 2) | Baseline (8:00, 10:00, 16:00); Day 8 (8:00, 10:00, 16:00); Day 15 (8:00, 10:00, 16:00); Day 29 (8:00, 10:00, 16:00)
  Intraocular pressure (IOP) will be measured with a Goldmann tonometer. The baseline mean diurnal IOP will be calculated as the average of the three baseline measurements. Baseline is defined as the last visit prior to initiation of treatment.
Mean percent change from baseline mean diurnal IOP at each post-treatment timepoint (Stage 2) | Baseline (8:00, 10:00, 16:00); Day 8 (8:00, 10:00, 16:00); Day 15 (8:00, 10:00, 16:00); Day 29 (8:00, 10:00, 16:00)
  Intraocular pressure (IOP) will be measured with a Goldmann tonometer. The baseline mean diurnal IOP will be calculated as the average of the three baseline measurements. Baseline is defined as the last visit prior to initiation of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Pharma, Study Director — Alcon Research, LLC
Locations (12):
- United States (12):
  - Orange County Ophthalmology Medical Group, Garden Grove, California
  - United Medical Research Institute, Inglewood, California
  - Eye Research Foundation, Newport Beach, California
  - North Bay Eye Associates, Petaluma, California
  - Eye Center of Northern Colorado, PC, Fort Collins, Colorado
  - Coastal Research Associates, Roswell, Georgia
  - Rochester Ophthalmological Group, Rochester, New York
  - James D. Branch Ophthalmology, Winston-Salem, North Carolina
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - University Eye Specialists, Maryville, Tennessee
  - Total Eye Care PA, Memphis, Tennessee
  - Piedmont Eye Center, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No